CLINICAL TRIAL: NCT01784185
Title: Development and Evaluation of Clinical Utility of Virtual Bronchoscopy (VB)-Based System for Bronchoscopic Navigation, Mediastinal Mapping and Transbronchial Aspiration of Mediastinal Lesions.
Brief Title: Virtual Bronchoscopy (VB) vs. Endobronchial Ultrasound (EBUS) Guided Mediastinal Sampling
Acronym: VB/EBUS-TBNA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Warsaw University of Technology (Other)
Responsible Party: Principal Investigator, Rafał Krenke, MD, PhD, Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: IPU-DIMPA-WUM12(1)
Record Dates: First submitted 2013-01-24; First posted 2013-02-05 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Lung Cancer,; Mediastinal Tumors,; Lymphomas,; Sarcoidosis,
Keywords: EBUS guided transbronchial needle aspiration (EBUS-TBNA); virtual bronchoscopy (VB); VB guided transbronchial needle aspiration VB-TBNA); mediastinal sampling; transbronchial needle aspiration (TBNA)
MeSH Terms: conditions — Lung Neoplasms; Lymphoma; Sarcoidosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- virtual bronchoscopy guided transbronchial needle aspiration (Experimental): virtual bronchoscopy guided transbronchial needle aspiration (VB-TBNA)(experimental method) and EBUS-TBNA (reference method) are performed in the same diagnostic session
  Interventions: Procedure: virtual bronchoscopy guided transbronchial needle aspiration; Procedure: endobronchial ultrasound guided transbronchial needle aspiration

INTERVENTIONS:
Procedure: virtual bronchoscopy guided transbronchial needle aspiration
  Other Names: VB-TBNA
Procedure: endobronchial ultrasound guided transbronchial needle aspiration — endobronchial ultrasound guided transbronchial needle aspiration (EBUS-TBNA) of mediastinal lesions
  Other Names: EBUS-TBNA

SUMMARY:
The study has been designed to evaluate the clinical application of the new virtual bronchoscopy (VB) -based system for transbronchial sampling of the mediastinal masses or enlarged lymph nodes. The software uses data from thorax CT scan and enables airway segmentation and reconstruction simultaneously with predefined mediastinal targets. The most suitable sites for transbronchial needle aspiration are displayed on the internal surface of the airways showed in VB mode.

The diagnostic yield of the new system-assisted TBNA will be compared to the reference method (EBUS-TBNA). The study group includes patients with mediastinal mass or lymph node enlargement in whom diagnostic bronchoscopy and TBNA can be applied as diagnostic methods. Both, virtual bronchoscopy guided transbronchial needle aspiration (VB-TBNA) and EBUS-TBNA of the mediastinal targets are performed during the same diagnostic bronchoscopy. Cytologic material from VB-TBNA and EBUS-TBNA is evaluated by two independent pathologists blinded to the method used to obtain the sample. Diagnostic yield and adequacy of aspirates obtained with the two methods will be assessed and compared.

ELIGIBILITY:
Inclusion Criteria:

* provided informed consent
* mediastinal mass or lymph node enlargement that requires bronchoscopy and transbronchial sampling
* quality of the CT scan which allows bronchial tree and mediastinal target segmentation and reconstruction

Exclusion Criteria:

* Age below 18 years
* known contraindications for bronchoscopy and/or mediastinal sampling, e.g. coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-02 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Adequacy of cytologic specimens collected by VB-TBNA vs. EBUS-TBNA | Approximately five days after the procedure, when the results of the cytological examination will be available
  Comparison of the quality and adequacy of the cytologic specimens (in terms of lymphocyte percentage, the presence of neoplastic cells and dust-laden macrophages) collected by VB-TBNA vs. EBUS-TBNA in patients with mediastinal mass or mediastinal lymph node enlargement

SECONDARY OUTCOMES:
Diagnostic accuracy of VB-TBNA vs. EBUS-TBNA - the number (and percentage) of cytologic specimens containing diagnostic material (neoplastic cells, granulomas) | up to 8 months
  Comparison of the diagnostic accuracy of VB-TBNA vs. EBUS-TBNA (in terms of number of cytologic specimens containing diagnostic material e.g. neoplastic cells, granulomas) in patients with mediastinal mass or mediastinal lymph node enlargement. Also the number of patients in whom the specific diagnosis could be established by VB-TBNA vs EBUS-TBNA.

OTHER OUTCOMES:
Number of patients with local complications of VB-TBNA | During VB-TBNA and EBUS-TBNA procedure
  Number of patients in whom large mediastinal vessels would be injured when performing VB-TBNA will be compared with respective number of patients with EBUS-TBNA associated large vessel injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Pneumonology and Allergology, Medical University of Warsaw, Warsaw, Poland